CLINICAL TRIAL: NCT02137265
Title: A Randomized, Double-blind, Placebo-controlled Trial of Clomiphene Citrate of Clomiphene Citrate in Hypoandrogenism and Azoospermia
Brief Title: Assessing the Efficacy of Clomiphene Citrate in Patients With Azoospermia and Hypoandrogenism
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding obtained
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Dr. Craig Niederberger, Clarence C. Saelhof Professor and Head, Department of Urology, UIC College of Medicine, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014-0343
Record Dates: First submitted 2014-05-09; First posted 2014-05-13 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Non Obstructive Azoospermia; Hypogonadism
Keywords: Azoospermia; Hypogonadism; Clomiphene
MeSH Terms: conditions — Hypogonadism; Azoospermia | interventions — Clomiphene

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clomiphene citrate (Active Comparator): Clomiphene citrate 50 mg daily during 4-6 months
  Interventions: Drug: Clomiphene
- Placebo (Placebo Comparator): Placebo (1 pill daily) during 4-6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clomiphene — Clomiphene citrate 50 mg orally daily
  Other Names: Clomid; Serophene
  Arms: Clomiphene citrate
Drug: Placebo — One pill every other day
  Other Names: control
  Arms: Placebo

SUMMARY:
Hypothesis: Prescribed clomiphene citrate to azoospermic patients with hypoandrogenism could improve the sperm retrieval in either fresh sperm or after surgical sperm extraction.

DETAILED DESCRIPTION:
Hypogonadism (low testosterone level) is frequently observed in men presenting with non obstructive azoospermia. Controversy exists regarding the efficacy of preoperative hormonal manipulation in patients with hypogonadism. However, it is possible that hormonal therapy increases intra-testicular testosterone levels, and with a rise in serum testosterone, sperm production and surgical success with microTESE improve.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old.
* Man seeking fertility treatment.
* Azoospermia confirmed in at least 2 semen analyses with centrifugation.
* Testosterone <300 ng/dL and Bioavailable Testosterone<156 ng/dL.

Exclusion Criteria:

* Presence of genetic disorders: Y chromosome deletions or abnormal karyotypes.
* Luteinizing hormone (LH) >25 IU/mL.
* Estradiol > 40 ng/dL.
* Hypogonadotropic hypogonadism (LH <2 IU/mL and Follicle Stimulating Hormone (FSH) <1 IU/mL).
* Obstructive azoospermia (FSH <7.6 IU/mL plus testicle longitudinally axis >4.6 cm or bilateral absence of vas deferens or surgical history of vasectomy).
* Clinical varicocele (palpable or visible in physical exam)
* Previous history of cryptorchidism.
* Use of chemotherapy, testosterone, or anti-androgen in the last two years. Partner >40 years or female factor infertility associated.
* Contraindications to clomiphene use: depression, heart and liver impairment, uncontrolled thyroid/adrenal dysfunction, organic intracranial lesions.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2020-10 (Actual); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Presence of sperm in the ejaculated or in the microsurgical testicular Sperm extraction (microTESE) | After four months of clomiphene treatment
Epigenetic modifications | After four months of clomiphene treatment

SECONDARY OUTCOMES:
Testosterone levels and Bioavailable Testosterone levels | After two weeks and four months with clomiphene treatment

CONTACTS AND LOCATIONS:
Overall Officials: Saturnino Luján, MD, PhD, Study Chair — University of Valencia
Locations (1):
- University of Valencia, Valencia, Province of Valencia, Spain

REFERENCES:
- [Result] Hussein A, Ozgok Y, Ross L, Niederberger C. Clomiphene administration for cases of nonobstructive azoospermia: a multicenter study. J Androl. 2005 Nov-Dec;26(6):787-91; discussion 792-3. doi: 10.2164/jandrol.04180. PMID 16291975
- [Result] Hussein A, Ozgok Y, Ross L, Rao P, Niederberger C. Optimization of spermatogenesis-regulating hormones in patients with non-obstructive azoospermia and its impact on sperm retrieval: a multicentre study. BJU Int. 2013 Mar;111(3 Pt B):E110-4. doi: 10.1111/j.1464-410X.2012.11485.x. Epub 2012 Sep 7. PMID 22958644